CLINICAL TRIAL: NCT02675725
Title: Kinetics of the Sublingual Microcirculation During the Treatment of a Postoperative Shock
Brief Title: Kinetics of the Sublingual Microcirculation During Fluid Bolus
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Gerke Veenstra, MD, Frisius Medisch Centrum
Other Study IDs: nWMO 128
Record Dates: First submitted 2016-01-08; First posted 2016-02-05 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2017-03

CONDITIONS: Surgery; Hypovolemic Shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post cardiac surgery: Patients after cardiac surgery with signs of decreased organ perfusion and the need of fluid therapy.
  Interventions: Device: Measurement of sublingual microcirculation with Cytocam-IDF camera

INTERVENTIONS:
Device: Measurement of sublingual microcirculation with Cytocam-IDF camera — The normal treatment of a post-cardiac surgery patient is fluid bolus by indication. This indications are hypotension, hyperlactataemia, tachycardia or decreased urine production. This fluid bolus is 250 ml crystalloids in 15 minutes.
  When this fluid bolus will be given, the investigators will observe the sublingual microcirculation and measure the red blood cell velocity and total vessel density on one spot for 20 minutes.

SUMMARY:
Fluid therapy is one of the cornerstones of the treatment of organ failure. The investigators assume that fluid bolus will increase the delivery of oxygen to the cells and resolve the shock.

The purpose of this study is to asses kinetics of the sublingual microcirculation in one place during a fluid bolus. It is expected that fluid therapy after normalization of the red blood cell flow velocity in the microcirculation will result in a decrease in capillary density through the formation of edema in the tissues. This can be considered to be the tipping of potentially beneficial to deleterious effects of fluid therapy.

After cardiac surgery patient will be transferred to the ICU for further stabilisation. Within specific indications the patient will receive a fluid bolus, these indications are hypotension, hyperlactataemia, tachycardia or decreased urine production. The fluid bolus will be 250 ml crystalloids in 15 minutes. The investigators will observe the sublingual microcirculation during this fluid bolus. To asses the red blood cell velocity and capillary vessel density on one spot during this fluid bolus.

DETAILED DESCRIPTION:
Fluid therapy is one of the cornerstones of the treatment of organ failure. The investigators assume that a fluid bolus will increase the delivery of oxygen to the cells and resolve the shock. The evaluation of this treatment is done by clinical signs of organ perfusion en (little used) invasive hemodynamic monitoring. Previous research suggests that in-vivo microscopy of the microcirculation can be of importance to determine the type of shock and the reaction on treatment on tissue level.

Evaluation of the microcirculation was done by measuring red blood cell velocity on three different sites in the sublingual region. This was necessary in order to take heterogeneity into account, it was very hard to fix the camera on one spot during the observation period.

The purpose of this study is to asses kinetics of the sublingual microcirculation in one place during a fluid bolus. The great advantage is that the recordings before and after fluid therapy can be compared with each other as paired data, wherein the subject is its own control. By choosing a time interval that is long enough for the observation of the changes, but short enough for manual fixing of the camera, it seems possible to serve both purposes (15-30 minutes). This seems crucial now because both red blood cell flow as capillary density will be measured. It is expected that fluid therapy after normalization of the red blood cell flow velocity in the microcirculation will result in a decrease in capillary density through the formation of edema in the tissues. This can be considered to be the tipping of potentially beneficial to deleterious effects of fluid therapy.

After cardiac surgery patient will be transferred to the ICU for further stabilisation. Within specific indications the patient will receive a fluid bolus, these indications are hypotension, hyperlactataemia, tachycardia or decreased urine production. The fluid bolus will be 250 ml crystalloids in 15 minutes. The investigators will observe the sublingual microcirculation during this fluid bolus. To asses the red blood cell velocity and capillary vessel density on one spot during this fluid bolus.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* post-cardiac surgery and need for fluid therapy

Exclusion Criteria:

* recent maxillofacial surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postoperative cardiac surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Change in Red blood cell velocity | before start fluid bolus, 5 min, 10 min, 15 min, 20 min after the start of the fluid bolus
  Measuring red blood cell velocity by using the microcirculatory blood flow index by eye-balling, (0: no flow; 1: stop-and-go; 2: sluggish; 3: normal flow)

SECONDARY OUTCOMES:
Change in Capillary vessel density | before start fluid bolus, 5 min, 10 min, 15 min, 20 min after the start of the fluid bolus
  Offline analysis of the images made on known time points will provide a total vessel density change during the fluid bolus. Total vessel density: area of vessels divided by the total area of the image, mm/mm2.

CONTACTS AND LOCATIONS:
Overall Officials: E.C. Boerma, MD-PhD, Principal Investigator — Frisius Medisch Centrum
Locations (1):
- Medical Centre Leeuwarden, Leeuwarden, Provincie Friesland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pranskunas A, Koopmans M, Koetsier PM, Pilvinis V, Boerma EC. Microcirculatory blood flow as a tool to select ICU patients eligible for fluid therapy. Intensive Care Med. 2013 Apr;39(4):612-9. doi: 10.1007/s00134-012-2793-8. Epub 2012 Dec 20. PMID 23263029
- [Background] Veenstra G, Ince C, Boerma EC. Direct markers of organ perfusion to guide fluid therapy: when to start, when to stop. Best Pract Res Clin Anaesthesiol. 2014 Sep;28(3):217-26. doi: 10.1016/j.bpa.2014.06.002. Epub 2014 Jul 15. PMID 25208957
- [Background] van Genderen ME, Klijn E, Lima A, de Jonge J, Sleeswijk Visser S, Voorbeijtel J, Bakker J, van Bommel J. Microvascular perfusion as a target for fluid resuscitation in experimental circulatory shock. Crit Care Med. 2014 Feb;42(2):e96-e105. doi: 10.1097/CCM.0b013e3182a63fbf. PMID 24158169
- [Background] Xu J, Ma L, Sun S, Lu X, Wu X, Li Z, Tang W. Fluid resuscitation guided by sublingual partial pressure of carbon dioxide during hemorrhagic shock in a porcine model. Shock. 2013 Apr;39(4):361-5. doi: 10.1097/SHK.0b013e31828936aa. PMID 23364438
- [Background] Ince C. The rationale for microcirculatory guided fluid therapy. Curr Opin Crit Care. 2014 Jun;20(3):301-8. doi: 10.1097/MCC.0000000000000091. PMID 24758985